CLINICAL TRIAL: NCT02007226
Title: Coronary Artery Calcification (CAC) Score and Risk Factors for Coronary Artery Disease in Persons With Spinal Cord Injury(SCI)
Brief Title: Coronary Artery Calcification Score and Risk Factors for Coronary Artery Disease in Persons With Spinal Cord Injury
Acronym: CAC
Status: Completed | Type: Observational
Sponsor: James J. Peters Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, William A. Bauman, M.D., Director: SCI Research Center, James J. Peters Veterans Affairs Medical Center
Other Study IDs: BAU-11-075
Record Dates: First submitted 2012-12-14; First posted 2013-12-10 (Estimated); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Spinal Cord Injury
Keywords: Coronary Heart Disease; spinal cord injury; risk factor; postprandial lipemia
MeSH Terms: conditions — Spinal Cord Injuries; Coronary Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum and Plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Spinal Cord Injury: Chronic SCI (Duration of Injury >5 years)

SUMMARY:
Although conventional risk factors for coronary heart disease (CHD) have been identified and routinely used to determine risk for CHD in the general population, a systematic approach to determine population-specific risk for CHD has not been performed prospectively in those with SCI. CHD is a leading cause of death in spinal cord injury, occurring at younger ages than in the able-bodied population. Conventional risk factors for CHD are high serum concentrations of low-density lipoprotein (LDL), low serum concentrations of high-density lipoprotein (HDL), diabetes mellitus (DM), positive smoking history, and positive family history of premature CHD.

Coronary Artery calcification (CAC) is a commonly occurring phenomenon that does not necessarily indicate significant obstructive disease. Studies have shown that a strong association exists between coronary calcification and coronary heart disease. The purpose of this study is to compare the CAC scores in persons with SCI with a historical control group of able-bodied persons from a national data base who will be matched for conventional risk factors for coronary artery disease (CAD) and to determine the relationship between CAC scores and conventional and emerging risk factors for CAD. Additionally, postprandial lipemic (elevated levels of lipids following ingestion of food) responses among individuals with SCI and control subjects will be compared, as well as the response of inflammatory markers following a high fat meal. Participants will only be tested once for these parameters.

DETAILED DESCRIPTION:
The early identification of individuals at high risk for development of CVD has been a challenging and highly relevant pursuit for clinicians and epidemiologists. The clinical significance of early identification of CAD becomes apparent because several of the cardiac risk factors are modifiable. Numerous studies have been performed to identify risk factors for CVD. These studies resulted in clinical guidelines for identification and risk reduction for CVD, currently summarized in the Third Report of the Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults: Adult Treatment Panel (ATP III). ATP III identifies five major risk factors for CVD: hyperlipidemia, hypertension, current smoking, abdominal obesity, and diabetes; individuals with two or more risk factors are considered at increased risk, although this recommendation may be changed to one risk factor in the upcoming ATP IV.

From a clinical perspective however, shortcomings in the prognostic value of the current conventional risk factors are becoming increasingly apparent. Retrospective reviews of large cohort studies and clinical trials conducted in the general population have found that ≥1 major conventional risk factor was present in 90% of patients who had diagnosed CAD. However, approximately 70% of subjects with established risk did not develop an event related to CAD during a 21-30 year follow-up period. These findings suggest that major predictors of CAD risk, although up to 90% sensitive, may be just 30% specific.

In persons with chronic SCI (> 1 year), cardiovascular disease (CVD) is a leading cause of mortality, as it is in the general population. Compared to the general population, CVD-related morbidity in persons with SCI, specifically CAD, occurs earlier in life and is more prevalent. Based on this knowledge, the need for appropriate risk stratification in SCI population becomes apparent. Existing tools do not take into account specific consequences of SCI, possibly underestimating the actual risk for CVD. For example, most of the risk factor algorithms incorporate HDL cholesterol into their equations to determine CAD risk, with a cutoff level of HDL cholesterol below which the general population is at a heightened risk for disease. Such an approach does not factor in the severity of depression of HDL cholesterol. It is appreciated that the morbidity risk ratio for CAD in men rises above unity at an HDL cholesterol <40 mg/dL, and the risk continues to rise in a linear fashion as the values for the lipid moiety decrease. In individuals with SCI, HDL cholesterol levels may be markedly depressed, with higher, more complete lesions having the lowest values. Thus, individuals with SCI will have additional risk for CAD based on extremely depressed values of HDL cholesterol that are not captured by conventional categorization. In addition, higher cord lesions (above thoracic level six) are frequently hypotensive, activating the renin-angiotensin axis in an attempt to maintain normotension. Elevated levels of angiotension are appreciated be atherogenic. Once again, this pathophysiologic condition-that is, hypotension and elevated angiotensin levels- is not captured by conventional risk factor paradigms. Because of these considerations, as well as the extreme immobilization of SCI that may independently confer additional CAD risk, the use of conventional risk assessment tools in this population is fraught with obvious difficulty and potential error. For years, the need for development of new non-conventional assessment tools has been recognized in the able-bodied population, and the need for a more reliable vehicle to identify individuals at heightened risk is even more the case in individuals with SCI.

The predictive value of emerging risk factors has been studied in an attempt to increase both the sensitivity and specificity of the identification of individuals at heightened risk of CAD, and thus to improve early diagnoses and result in the appropriate institution of efficacious risk modification approaches. Abdominal fat, inflammatory biomarkers, CAC, arterial stiffness, increased C-reactive protein (CRP), vitamins and antioxidant deficiency, endothelial dysfunction, increased arterial intima media thickness (IMT), triglyceride response to fat load, and genetic factors have been extensively studied as potential predictors of increased risk for CAD in the general population.

Among the non-conventional approaches, measurement of CAC scores has been most promising. CAC is highly specific to the atherosclerosis and is thought to develop late in its pathophysiology, reflecting a chronic plaque burden. CAC has been used in the global CVD risk stratification of asymptomatic patients to identify additional risk among those with a seemingly low-risk; the additional predictive value of CAC for CAD risk was greater than that provided by the conventional risk factors, regardless of racial or ethnic considerations. The higher the CAC score, the greater the prevalence of myocardial perfusion abnormalities associated with obstructive CAD and risk of death or myocardial infarction within 3 to 5 years. Approximately two-thirds of persons with SCI have intermediate risk for CAD; evidence suggests that many have silent CAD. Of note, and somewhat troubling, in reports in symptomatic individuals without CAC, 16-24% have obstructive CAD, an observation corroborated by the finding that approximately 20% of occluded vessels may not have detectable calcification.

ELIGIBILITY:
Inclusion Criteria:

* Males 45-75 years old with at least 5 yrs of SCI
* Females 50-75 years old with at least 5 yrs of SCI; females 40-50 years old with at least 10 yrs of SCI;
* Stable SCI (regardless of level of lesion or completeness of injury).
* Ability to sign consent form.

For Optional Fat Meal Test Only

* Must have completed initial risk factor assessment as previously described.

Exclusion Criteria:

* Acute medical illness;
* Pregnancy;
* Chronic debilitating disease (i.e., severe pulmonary disease, stage IV pressure ulcers, etc.);
* Atrial fibrillation;
* History of percutaneous coronary angiography with stent placement.

For Optional Fat Meal Test Only:

* Known diabetes;
* Lactose-intolerance or dairy allergy;
* Allergy to chocolate.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from hospital clinics, through advertisements, and referral from primary care physicians
Sampling Method: Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2020-04 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Coronary heart disease risk factors | Testing will be performed at day 1 for all parameters
  The relationship of coronary artery calcification (CAC) with conventional risk factors (cigarette smoking, hypertension, low high density lipoprotein(HDL) cholesterol, diabetes) and nonconventional risk factors (abdominal fat, inflammatory biomarkers, arterial stiffness, intima media thickness of carotid artery) is being tested to determine the prevalence and severity of coronary artery calcification (CAC) score of SCI individuals with age, gender and ethnically matched controls.

SECONDARY OUTCOMES:
Postprandial lipemic response to a high fat meal(1.3 gm/kg body weight) | Single fat meal challenge test will be performed at day 1.
  To determine the postprandial lipemic response to fat load in persons with SCI and to correlate these parameters to other risk factors for CAD and CAC score.

CONTACTS AND LOCATIONS:
Overall Officials: William A Bauman, MD, Principal Investigator — James J. Peters Veterans Affairs Medical Center
Locations (2):
- United States (2):
  - Kessler Institute for Rehabilitation, West Orange, New Jersey
  - James J Peters VA Medical Center, The Bronx, New York

REFERENCES:
- [Background] Emmons RR, Garber CE, Cirnigliaro CM, Moyer JM, Kirshblum SC, Galea MD, Spungen AM, Bauman WA. The influence of visceral fat on the postprandial lipemic response in men with paraplegia. J Am Coll Nutr. 2010 Oct;29(5):476-81. doi: 10.1080/07315724.2010.10719884. PMID 21504974
- [Background] Bauman WA, Spungen AM. Carbohydrate and lipid metabolism in chronic spinal cord injury. J Spinal Cord Med. 2001 Winter;24(4):266-77. doi: 10.1080/10790268.2001.11753584. PMID 11944785
- [Background] Bauman WA, Spungen AM. Metabolic changes in persons after spinal cord injury. Phys Med Rehabil Clin N Am. 2000 Feb;11(1):109-40. PMID 10680161
- [Background] Bauman WA, Spungen AM. Disorders of carbohydrate and lipid metabolism in veterans with paraplegia or quadriplegia: a model of premature aging. Metabolism. 1994 Jun;43(6):749-56. doi: 10.1016/0026-0495(94)90126-0. PMID 8201966
- [Background] Bauman WA, Spungen AM, Raza M, Rothstein J, Zhang RL, Zhong YG, Tsuruta M, Shahidi R, Pierson RN Jr, Wang J, et al. Coronary artery disease: metabolic risk factors and latent disease in individuals with paraplegia. Mt Sinai J Med. 1992 Mar;59(2):163-8. PMID 1574072
- [Derived] McCauley LS, Ghatas MP, Sumrell RM, Cirnigliaro CM, Kirshblum SC, Bauman WA, Gorgey AS. Measurement of Visceral Adipose Tissue in Persons With Spinal Cord Injury by Magnetic Resonance Imaging and Dual X-Ray Absorptiometry: Generation and Application of a Predictive Equation. J Clin Densitom. 2020 Jan-Mar;23(1):63-72. doi: 10.1016/j.jocd.2018.12.003. Epub 2018 Dec 15. PMID 30638769